CLINICAL TRIAL: NCT03578107
Title: Improve Acute Reperfusion Treatment Quality for Stroke in China
Brief Title: Improve Acute Reperfusion Treatment Quality for Stroke in China, IMPROVE: Stroke Care in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Yongjun Wang, Executive Vice-President, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: KY 2018-044-01
Record Dates: First submitted 2018-06-24; First posted 2018-07-05 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Ischemic Stroke
Keywords: acute ischemic stroke; IV-tPA; endovascular treatment; intervention
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Improvement intervention1 (Other): receive the following improvement intervention for 18 months：
  Interventions: Behavioral: improvement of quality of stroke care
- Improvement intervention2 (Other): receive the following improvement intervention for 12 months：
  Interventions: Behavioral: improvement of quality of stroke care
- Improvement intervention3 (Other): receive the following improvement intervention for 6 months：
  Interventions: Behavioral: improvement of quality of stroke care

INTERVENTIONS:
Behavioral: improvement of quality of stroke care — 1. hospital tool kits for quality improvement of reperfusion therapy ;
  2. organizational stakeholder and opinion leader meetings;
  3. data monitoring and feedback reports；
  4. webinar for hospital teams

SUMMARY:
In order to bridge the great gaps, Chinese Stroke Association (CSA) and American Heart Association (AHA) sought to develop, conduct, and assess a multifaceted quality improvement intervention to increase the adherent rate of IV tPA and ET and improve 3-month clinical outcomes for these patients through our cluster-randomized stepped-wedge IMPROVE: Stroke in China trial.

ELIGIBILITY:
Inclusion Criteria:

Hospitals：

1. Voluntary.
2. Hospitals from CSCA.
3. Secondary or tertiary public hospitals with an emergency department and neurologic wards that receive patients with AIS.
4. Have a 24*7 on-call stroke team.
5. Have the capacity of IV rt-PA thrombolytic therapy or/and endovascular treatment.
6. Implement at least 10 patients' rt-PA or/and endovascular treatment during the last year.
7. Admit at least 5 patients of acute ischemic stroke within 24 hours after onset each month.
8. Have full desire to improve the procedure of treatment of acute ischemic stroke.
9. Have good cooperation among Neurology department, Emergency department, Interventional department, Neurosurgery department, Laboratory and Radiology department.

Patients： Patients who are ≥18 years old were eligible for inclusion if they presented with acute ischemic stroke diagnosed by CT and/or MRI and arrived at hospital within 6 hours after symptom onset.

Exclusion Criteria:

Hospitals：

1. Hospitals that can not comply with the protocol and finish the research.
2. Grade-one hospitals and non cerebral vascular disease specialized hospitals.
3. Hospitals involved in other stroke care quality improvement projects or relevant clinical trials.

Patients：

1）Patients refuse to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15895 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
The adherence rate of guidelines for IV-tPA and/or endovascular treatment in eligible patients. | participants will be followed for the duration of hospital stay, an expected average of 2 weeks

SECONDARY OUTCOMES:
proportional change of intravenous thrombolytic therapy in eligible patients 4.5h after the onset | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
proportional change of endovascular treatment in eligible patients 6h after the onset | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
time from arrival to hospitals to intravenous thrombolytic therapy | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
door-to-puncture time | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
in-hospital mortality | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
3-month disability（mRS≥3 ） | patients will be followed up at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang CJ, Gu HQ, Zong LX, Zhang XM, Zhou Q, Jiang Y, Li H, Meng X, Yang X, Wang M, Huo XC, Wangqin RQ, Bei YZ, Qi XH, Liu XY, Hu SQ, Wang ZM, Zhao XQ, Wang YL, Liu LP, Ma XD, Morgan L, Xian Y, Schwamm LH, Wang YJ, Li ZX; IMPROVE Stroke Care in China investigators. Effectiveness of a Quality Improvement Intervention on Reperfusion Treatment for Patients With Acute Ischemic Stroke: A Stepped-Wedge Cluster Randomized Clinical Trial. JAMA Netw Open. 2023 Jun 1;6(6):e2316465. doi: 10.1001/jamanetworkopen.2023.16465. PMID 37266940
- [Derived] Li Z, Wang C, Zhang X, Zong L, Zhou H, Gu H, Jiang Y, Pan Y, Meng X, Zhou Q, Zhao H, Yang X, Wang M, Xiong Y, Zhao X, Wang Y, Liu L, Ma X, Morgan L, Xian Y, Schwamm LH, Wang Y. Rationale and design of a stepped wedge cluster randomised trial to improve acute reperfusion treatment quality for stroke: IMPROVE stroke care in China. Stroke Vasc Neurol. 2022 Oct;7(5):451-456. doi: 10.1136/svn-2021-001461. Epub 2022 Mar 30. PMID 35354662